CLINICAL TRIAL: NCT02183441
Title: Relative Bioavailability of a Single Oral Dose of BI 1356 (5 mg) After Co-administration With Multiple Oral Doses of Ritonavir (200 mg Bid for 3 Days) Compared to the Bioavailability of a Single Oral Dose of BI 1356 (5 mg) Alone in Healthy Male Volunteers (an Open-label, Randomized, Two-way Crossover, Clinical Phase I Study)
Brief Title: Bioavailability of BI 1356 After Co-administration With Ritonavir Compared to the Bioavailability of BI 1356 Alone in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1218.31
Record Dates: First submitted 2014-07-04; First posted 2014-07-08 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Linagliptin; Ritonavir

ARMS (2):
- BI 1356 plus ritonavir (Experimental): Treatment A: 3 days of ritonavir, 1 day BI 1356
  Interventions: Drug: BI 1356; Drug: Ritonavir
- BI 1356 (Active Comparator): Treatment B: BI 1356 alone
  Interventions: Drug: BI 1356

INTERVENTIONS:
Drug: BI 1356
Drug: Ritonavir
  Other Names: Norvir®
  Arms: BI 1356 plus ritonavir

SUMMARY:
Study to investigate the effect of the P-gp and cytochrome P450 (CYP) 3A4 inhibitor ritonavir on the pharmacokinetics of BI 1356

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria: Based upon a complete medical history, including the physical examination, vital signs (blood pressure (BP), pulse rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory tests
* Age ≥ 18 and Age ≤ 50 years
* BMI ≥ 18.5 and BMI ≤ 29.9 kg/m2 (Body Mass Index)
* Signed and dated written informed consent prior to admission to the study in accordance with good clinical practice (GCP) and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
* Surgery of the gastrointestinal tract (except appendectomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections (e.g. HIV)
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than five half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial (especially unspecific inducing agents like St.John´s wort (Hypericum perforatum) or drugs which prolong the QT/QTc interval based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day) or inability to stop alcoholic beverages for 24 hours prior to dosing and up to the last sampling time point
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a QTc interval >450 ms)
* A history of additional risk factors for torsades de points (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)

Exclusion criteria specific for this study:

* Galactose intolerance
* Lactase deficiency
* Glucose-galactose-malabsorption

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
AUC0-24 (Area under the concentration-time curve of BI 1356 in plasma over the time interval from 0 to 24 hours) | up to 24 hours after start of treatment
Cmax (Maximum measured concentration of BI 1356 in plasma) | up to 96 hours after start of treatment

SECONDARY OUTCOMES:
AUC (Area under the concentration time curve of the analytes in plasma at different time points) | up to 96 hours after start of treatment
%AUCtz-∞ (Percentage of the extrapolated part of the area under the concentration time curve of the analytes in plasma from 0 to infinity) | up to 96 hours after start of treatment
tmax (Time from dosing to the maximum concentration of the analytes in plasma) | up to 96 hours after start of treatment
t1/2 (Terminal half-life of the analytes in plasma) | up to 96 hours after start of treatment
λz (Terminal rate constant of the analytes in plasma) | up to 96 hours after start of treatment
MRTpo (Mean residence time in the body after po administration of the analytes in plasma) | up to 96 hours after start of treatment
CL/F (Apparent clearance of BI 1356 in plasma after extravascular administration ) | up to 96 hours after start of treatment
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) of BI 1356 | up to 96 hours after start of treatment
Aet1-t2 (Amount of the analytes that is eliminated in urine from the time interval t1 to t2) | up to 24 hours after start of treatment
fet1-t2 (Fraction of BI 1356 excreted unchanged in urine from time point t1 to t2) | up to 24 hours after start of treatment
CLR,t1-t2 (Renal clearance of the analytes in plasma) | up to 24 hours after start of treatment
Cmax (Maximum measured concentration of CD 1750 in Plasma) | up to 96 hours after start of treatment
Number of patients with adverse events | up to 53 days